CLINICAL TRIAL: NCT04851600
Title: Adaptative Motor Behavior of Children With Unilateral Upper Limb Deficiency After Early Prosthetics.
Brief Title: Early Prosthetics in Children With Upper Limb Deficiency
Acronym: EARLIMB
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_24; 2021-A00108-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-02

CONDITIONS: Limb Deficiencies
Keywords: Unilateral congenital upper extremity deficiency; Early development; Motor skills; Rehabilitation of amputees; Upper extremity deficiency; Upper limb prosthesis; Adaptative behavior
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early introduction: Casting and delivery of a cosmetic upper limb prosthesis at 3-4 months old of age.
  Interventions: Device: prosthesis

INTERVENTIONS:
Device: prosthesis — Casting and delivery of a cosmetic upper limb prosthesis at 3-4 months old of age.

SUMMARY:
For children with congenital upper limb deficiency, introduction of the prosthesis is guided by clinical experience rather than by Evidence Based Medicine.

This study will assess early development in children with upper limb deficiency according to age at the introduction of the prosthesis.

This study will give new keys in these specific prosthesis cares.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child
* Aged from 1 month to 3 months and a half
* Placement of a prosthesis in a patient with isolated upper limb deficiency, type of congenital transverse unilateral amputation of the forearm segment
* Socially insured patient,
* Patient willing to comply with all study procedures and study duration
* Written informed consent from patient's legal guardians

Exclusion Criteria:

* Children with one or more high risk factors for neurodevelopmental disorders:

  * Very prematurity (<32 weeks of amenorrhea [SA])
  * Premature infants <37 WA with intrauterine growth retardation (IUGR) or low weight for gestational age (PAG) <3rd percentile or <- 2 SD for GA and sex according to national reference curves)
  * A presumed hypoxo-ischemic encephalopathy with an indication of therapeutic hypothermia
  * A perinatal arterial cerebrovascular accident (AVC) (diagnosed between the 20th week of fetal life and the 28th day of life including in premature newborns).
  * Cerebral growth anomalies: microcephaly with cranial perimeter <- 2 SD at birth verified secondarily or macrocephaly> + 3 SD for the term (persisting after a second measurement).
  * A family history of severe first-degree neurodevelopmental disorder (brother or sister or parent)
  * Symptomatic congenital cytomegalovirus infections and other infectious fetopathies: toxoplasmosis, Zika, rubella, etc.
  * Bacterial and viral herpetic meningoencephalitis
  * Complex congenital heart disease operated on: transposition of the large vessels; left ventricular hypoplastic syndrome.
  * Perinatal exposure to a major toxicant: certain antiepileptics (sodium valproate); severe exposure to alcohol and / or with signs of fetal disease.
  * Major, prolonged and repeated surgery (cardiac, cerebral, abdominal, thoracic).
* Exclusion of all deficiency forming part of a polymalformative, vascular syndrome (Poland syndrome), genetic cause ...
* Exclusion of all other forms of agenesis (bilateral, longitudinal, persistence of hand remains),
* Refusal of consent from one or both parents

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child with unilateral upper limb agenesis
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales version II Motor skills Domain score Motor skills Domain score | at 24 months old

SECONDARY OUTCOMES:
Assisting Hand Assessment | at 3 years old
Communication Domain Score | at 9 months old , at 24 months old
Daily living skills Domain Score at 9 and 24 months old | at 9 months old , at 24 months old, at 3 years old
Socialization Domain score | at 9 months old , at 24 months old, at 3 years old
Motor skills Domain score | at 9 months old

CONTACTS AND LOCATIONS:
Overall Officials: Alice TAQUET, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Ssr Pediatrique Marc Sautelet, Villeneuve-d'Ascq, France